CLINICAL TRIAL: NCT02735772
Title: Transobturator Approach for Paravaginal Repair a New Approach
Brief Title: Transobturator Approach for Paravaginal Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Ahmed Saaid, Dr.Hamdy Ahmed, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVRNA
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Intervention Model Description: All Patients included in the study will undergo repair of paravaginal defect using tge new technique described in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cystocele (Other): Arm: Patients with paravaginal defect cystocele
  Intervention: transobturator approach for paravaginal repair
  Interventions: Procedure: transobturator approach for paravaginal repair

INTERVENTIONS:
Procedure: transobturator approach for paravaginal repair — using TOT needle to apply suturs to white line

SUMMARY:
A new technique for Applying sutures to the white line in paravaginal repair.

DETAILED DESCRIPTION:
A new trial for transobturator repair of the paravaginal defect.

ELIGIBILITY:
Inclusion Criteria:

* paravaginal defect cystocele
* midline and paravaginal defect cystocele

Exclusion Criteria:

* uterine descent
* previous cystocele surgery

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
success rate | 6 months
  Evaluation of the postoperative degree of anterior vaginal wall descent using pelvic organ prolapse quantitative system

SECONDARY OUTCOMES:
lateral vaginal fornices elevation | 3 month
  test is negative means success
Operative time | 1 day
  Operative time
Intraoperative blood loss | 1 day
  Blood loss during the operative procedure
Complications rate | 1 week
  Intraoperative and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Hazem SH Samoor, Professor, Study Chair — Ain Shams Universty
Locations (1):
- Urogynecology Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No